CLINICAL TRIAL: NCT01494727
Title: A Randomized, Open-label, Single Dose, Two-way Crossover Clinical Trial to Compare the Safety, Pharmacokinetic Profiles of CJ Amlodipine/Valsartan 10/160mg Tablet and Novartis Exforge 10/160mg Tablet After a Single Oral Administration in Healthy Male Volunteers
Brief Title: Phase I Study to Compare the Safety, Pharmacokinetic Profiles of CJ Amlodipine/Valsartan 10/160mg and Novartis Exforge 10/160mg
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_AMV_101
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Healthy
Keywords: Safety; Pharmacokinetics
MeSH Terms: interventions — Valsartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CJ Amlodipine/Valsartan 10/160mg (Experimental)
  Interventions: Drug: CJ Amlodipine/Valsartan 10/160mg
- Novartis Exforge 10/160mg (Active Comparator)
  Interventions: Drug: Novartis Exforge 10/160mg

INTERVENTIONS:
Drug: CJ Amlodipine/Valsartan 10/160mg — single dose
  Arms: CJ Amlodipine/Valsartan 10/160mg
Drug: Novartis Exforge 10/160mg — single dose
  Arms: Novartis Exforge 10/160mg

SUMMARY:
The objectives of this study are:

* To compare the safety profile of CJ Amlodipine/Valsartan 10/160mg and Novartis Exforge 10/160mg after a single oral administration in healthy male volunteers
* To compare the pharmacokinetic profile of CJ Amlodipine/Valsartan 10/160mg and Novartis Exforge 10/160mg after a single oral administration in healthy male volunteers

ELIGIBILITY:
Inclusion Criteria:

* Male volunteers in the age between 20 and 45 years old
* Body Mass Index (BMI) in the range of 19 to 27 kg/m2

Exclusion Criteria:

* History of allergy or sensitivity to any drug, including amlodipine or valsartan
* History of clinically significant hepatic, renal, gastrointestinal, neurology, pulmonary, endocrine, musculoskeletal, hematologic, oncologic, psychiatric, especially cardiovascular disease
* History of surgery except or gastrointestinal diseases which might significantly change absorption of medicines
* Hypotension (Systolic Blood Pressure(SBP) ≤ 100 mmHg or Diastolic Blood Pressure(DBP) ≤ 65 mmHg)
* Hypertension (SBP ≥ 150 mmHg or DBP ≥ 95 mmHg)
* Clinical laboratory test values are outside the accepted normal range

  * Aspartate Transaminase(AST) or Alanine Transaminase(ALT) > 1.25 times to normal range
  * Total bilirubin > 1.25 times to normal range
* Positive for Hepatitis B Virus surface Antigen(HBsAg), Hepatitis C Virus Antibody(HCVAb) or Human Immunodeficiency Virus Antibody(HIVAb)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea